CLINICAL TRIAL: NCT04786210
Title: A Prospective Triple-Blinded Single-Center Study of Laser-Assisted 5-Fluorouracil Versus Laser-Assisted Corticosteroid Treatment for Keloids
Brief Title: Treatment of Keloids With Fractional Erbium Laser-Assisted 5-Fluorouracil Versus Laser-Assisted Corticosteroid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-01172
Record Dates: First submitted 2021-01-25; First posted 2021-03-08 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Keloid Scar
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Site A of keloid scar (Experimental): One half of keloid scarring on a single subject
  Interventions: Combination Product: Fractional erbium:YAG-assisted drug delivery of 5-fluorouracil
- Site B of keloid scar (Experimental): One half of keloid scarring on a single subject
  Interventions: Combination Product: Fractional erbium:YAG-assisted drug delivery of triamcinolone acetonide

INTERVENTIONS:
Combination Product: Fractional erbium:YAG-assisted drug delivery of 5-fluorouracil — Split-scar fractional ablative erbium laser-assisted delivery of 50mg/mL of 5-fluorouracil solution to one half of the scar (4 treatments)
  Arms: Site A of keloid scar
Combination Product: Fractional erbium:YAG-assisted drug delivery of triamcinolone acetonide — Split-scar fractional ablative erbium laser-assisted delivery of 10 mg/mL of triamcinolone acetonide solution to the other half of the scar (4 treatments)
  Arms: Site B of keloid scar

SUMMARY:
This is a split-scar study with a target sample size of 20. There are two interventions: fractional erbium:YAG-assisted drug delivery of 5-fluorouracil and fractional erbium:YAG-assisted drug delivery of triamcinolone acetonide. Patients will undergo treatments in a series of 4 treatments at approximately 4 week ± 1 week intervals. Investigators will monitor for safety and continued benefit after the end of the interventional treatment.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-89
2. Has one large keloid scar or at least two similar but separate keloid scars
3. Keloid present for at least 1 year

Exclusion Criteria

1. Currently pregnant
2. Currently breastfeeding
3. Have taken oral retinoids within 6 months of study initiation
4. Has had keloid treatment within 1 month of study initiation
5. Has active infection at treatment site
6. Has active malignancy
7. Presence of pedunculated keloid(s) or keloid(s) that are judged to be best treated with surgical excision first
8. Hypertrophic scars
9. Known hypersensitivity to TAC or 5-FU
10. Chronic systemic corticosteroid or immunosuppressive medication use
11. Has intolerance to anesthesia
12. Has known connective tissue disease
13. Has known infectious disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Lee, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to nayoung.lee@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: halves of keloid scarring
Groups:
- Overall Study Population: One half of keloid scarring (Site A of keloid scar) on a single subject will be assigned to 5-FU: Split-scar fractional ablative erbium laser-assisted delivery of 50mg/mL of 5-fluorouracil (5-FU) solution to one half of the scar (4 treatments)
  The other half of keloid scarring (Site B of keloid scar) on a single subject will be assigned to TAC: Split-scar fractional ablative erbium laser-assisted delivery of 10 mg/mL of triamcinolone acetonide (TAC) solution to the other half of the scar (4 treatments).
Period: Overall Study
Arm/Group | Overall Study Population
Started | 19; 38 halves of keloid scarring
Received 5-fluorouracil (5-FU) | 19; 19 halves of keloid scarring
Received Triamcinolone Acetonide | 19; 19 halves of keloid scarring
Completed | 13; 26 halves of keloid scarring
Not Completed | 6; 12 halves of keloid scarring
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Population
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 36 [26 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient and Observer Scar Assessment Scale (POSAS) Score From Baseline to Final Visit
Description: POSAS has two components, the observer (physician) portion and the patient portion. The observer grades on a scale of 1 to 10, 10 being the worst scar imaginable, six measures: vascularity, pigmentation, thickness, relief, pliability and surface area. The patient answers six questions regarding the characteristics of the scar, with each question being on a scale of 1 to 10. The scores of each category are summed to get the total POSAS score, with 120 being the highest score and representing the worst scar and 12 being the lowest score.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Keloid scar
Groups:
- Site A of Keloid Scar - 5-FU: One half of keloid scarring on a single subject
  Fractional erbium:YAG-assisted drug delivery of 5-fluorouracil: Split-scar fractional ablative erbium laser-assisted delivery of 50mg/mL of 5-fluorouracil solution to one half of the scar (4 treatments)
- Site B of Keloid Scar - TAC: One half of keloid scarring on a single subject
  Fractional erbium:YAG-assisted drug delivery of triamcinolone acetonide: Split-scar fractional ablative erbium laser-assisted delivery of 10 mg/mL of triamcinolone acetonide solution to the other half of the scar (4 treatments)
Arm/Group | Site A of Keloid Scar - 5-FU | Site B of Keloid Scar - TAC
Number analyzed (Participants) | 13 | 13
Number analyzed (Keloid scar) | 13 | 13
score on a scale | -20 (8) | -20.6 (13.1)

2. Primary Outcome: Change in Modified Hamilton Score
Description: The Hamilton scale consists of 4 items with a score range of 0 to 14, where 14 represents more severe scarring.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Keloid scar
Arm/Group | Site A of Keloid Scar - 5-FU | Site B of Keloid Scar - TAC
Number analyzed (Participants) | 14 | 14
Number analyzed (Keloid scar) | 14 | 14
score on a scale | -0.88 (1.79) | -1.36 (1.21)

3. Secondary Outcome: Change in Scar Measurement From Baseline to Final Visit
Description: Scar measurement will be calculated as the total volume (length x width x height) in cm3 of the scar, or (length x width) in cm2 if the scars are flush with the surrounding skin scar surface.
Time Frame: Baseline, Week 16
Measure: Mean (Standard Deviation); unit: cm^3
Units Other Than Participants: Keloid scar
Arm/Group | Site A of Keloid Scar - 5-FU | Site B of Keloid Scar - TAC
Number analyzed (Participants) | 13 | 13
Number analyzed (Keloid scar) | 13 | 13
cm^3 | -368.7 (692.9) | -310.7 (626.7)

ADVERSE EVENTS:
Time Frame: Through study completion, on average 1 year.
Description: Systematic - At each visit subsequent to visit 1, a standard questionnaire of side effects was administered to participants (yielding 4 assessments for side effects per participant). All-cause mortality was not assessed in this study.
Arm/Group | Site A of Keloid Scar - 5-FU | Site B of Keloid Scar - TAC
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 12/19 | 12/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Site A of Keloid Scar - 5-FU (N=19) | Site B of Keloid Scar - TAC (N=19)
Bleeding at site (Skin and subcutaneous tissue disorders) | 1 | 0
Bruising at site (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling/edema at site (Skin and subcutaneous tissue disorders) | 3 | 1
Burning at site (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema of site (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperpigmentation of site (Skin and subcutaneous tissue disorders) | 9 | 3
Hypopigmentation of site (Skin and subcutaneous tissue disorders) | 2 | 0
Itching at site (Skin and subcutaneous tissue disorders) | 8 | 6
Pain at site (Skin and subcutaneous tissue disorders) | 4 | 4
Spreading/growth of scar (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04786210/Prot_SAP_000.pdf